CLINICAL TRIAL: NCT01806155
Title: Prevalence of Post-craniotomy Headache in Siriraj Hospital
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Sirilak Suksompong, Associate Professor, Mahidol University
Other Study IDs: 734/2555(EC2)
Record Dates: First submitted 2013-03-03; First posted 2013-03-07 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2013-08

CONDITIONS: Adult Brain Tumor; Headache
Keywords: craniotomy; headache; postoperative
MeSH Terms: conditions — Brain Neoplasms; Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Craniotomy: Patient undergoing major craniotomy

SUMMARY:
Headache after major craniotomy may be a problem in taking care of the patients. The investigators want to identify the incidence of headache after major craniotomy and also the risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing major craniotomy

Exclusion Criteria:

* emergency surgery or traumatic patients
* may need postoperative ventilatory support more than 2 days
* cannot communicate
* psychiatric patients
* chronic use of benzodiazepine or drug abuse
* cannot follow the treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient undergoing major craniotomy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-03 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
The incidence of headache after major craniotomy | 3 months
  By asking the patients about the symptoms

SECONDARY OUTCOMES:
risk factors of headache after major craniotomy such as sex, education | 3 months
  by collecting the patients data

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok, Thailand